CLINICAL TRIAL: NCT00581815
Title: Spectroscopy With Surface Coils and Decoupling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Columbia University (Other); University of Pennsylvania (Other); St. George's Hospital, London (Other); Royal Marsden NHS Foundation Trust (Other); University Medical Center Nijmegen (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 97-014
Record Dates: First submitted 2007-12-20; First posted 2007-12-28 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Adrenal Cortical Cancer; Brain Cancer; Breast Cancer; CNS Cancer; Colon Cancer; HEENT Cancer; Hodgkin's Disease; Kaposi's Sarcoma; Liver Cancer; Lung Cancer; Non-Hodgkin's Lymphoma; Ovarian Cancer; Pancreatic Cancer; Prostate Cancer; Rectal Cancer; Renal Cancer; Sarcoma; Squamous Cell Carcinoma; Thyroid Cancer
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms; Central Nervous System Neoplasms; Colonic Neoplasms; Hodgkin Disease; Sarcoma, Kaposi; Liver Neoplasms; Lung Neoplasms; Lymphoma, Non-Hodgkin; Ovarian Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Rectal Neoplasms; Kidney Neoplasms; Sarcoma; Carcinoma, Squamous Cell; Thyroid Neoplasms

ARMS (1):
- 1 (Experimental)
  Interventions: Device: Proton-decoupled 31P MRS at 1.5T; Device: 1H Spectroscopy at 1.5T and 3T

INTERVENTIONS:
Device: Proton-decoupled 31P MRS at 1.5T — The study will use a dual 1H-31P surface coil pair obtained from IGG Medical Advances, Milwaukee, WI. The coil pair consists of a fixed, 12 cm square 31P resonator co-mounted with a flexible two-loop proton coil. The P.I. and colleagues have used this device for approximately 10 years with no apparent ill effects
Device: 1H Spectroscopy at 1.5T and 3T — The study will use surface coils manufactured by commercial vendors. The pulse sequence programs to be used will be monitored automatically by the scanner to insure that SAR limits are not exceeded.

SUMMARY:
The purpose of this study is to obtain chemical information from part of your body without a biopsy. This is done using a technique called magnetic resonance spectroscopy (MRS) which is similar to magnetic resonance imaging (MRI) except that signals are detected from the chemicals (spectroscopy) naturally present in your body using radio waves. To receive this information from your body, small loops of wire (surface coils), placed near the tissue of interest, may be used to more effectively detect signals that come from the chemicals in your body. The investigators may use a second radio channel simultaneously, which will allow us to obtain greater chemical information (decoupling). The results may also help us to understand how this study can be used to help other patients with your condition.

DETAILED DESCRIPTION:
The investigators propose to use 1H spectroscopy or 1H decoupled 31P NMR spectroscopy to obtain biochemical information about tumor metabolism in patients, both before and after antineoplastic therapy. In healthy volunteers, normal tissue metabolism will also be studied. It is hypothesized that metabolic information may be of prognostic significance, or may be useful for timing of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have suspected or documented neoplastic disease, strongly suspected or established by physical examination, history or conventional histologic biochemical or imaging techniques, or have surgical or aspiration biopsy that will be used to establish a diagnosis
* Patients with obstructive jaundice, both from malignant and non-malignant disease, will be considered for the study
* Patients/volunteers must be clinically stable and not require cardiovascular monitoring
* Patients must be 6 years of age or older and be able to cooperate for an approximately 60 minute examination
* Volunteers must be 18 years of age or older

Exclusion Criteria:

* Inability to cooperate for an MR exam
* Contraindication to MR: Pacemaker, Aneurysmal clips Any ferrous metallic implants which could be deflected by the magnet, Metal implants in field of view, Pregnant women, OR Age and mental status wherein he/she is unable to cooperate for MR study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 582 (Actual)
Dates: Start 1997-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To obtain high resolution spectra from tumors using surface coils to improve sensitivity. | 2 years

SECONDARY OUTCOMES:
In some of these studies, to enhance our spectral resolution and obtain additional metabolic information, we propose to use decoupling, which will increase both signal quality (the signal to noise ratio) and spectral resolution. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Koutcher, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.mskcc.org